CLINICAL TRIAL: NCT07010458
Title: Advancing Acne Care - Clinical Trials Open for Patient Enrollment
Brief Title: Exploring Acne Treatments Through Clinical Research Participation
Status: Not yet recruiting | Type: Observational
Sponsor: Power Life Sciences Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 44519879
Record Dates: First submitted 2025-05-30; First posted 2025-06-08 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-05

CONDITIONS: Acne
Keywords: Acne
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to understand the lived experiences of acne patients enrolled in a related clinical trial testing a particular treatment. The primary focus will be on tracking trial adherence and dropout rates to enhance future research and care approaches, especially for underserved groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with acne.
* Aged ≥ 18 years old and ability to provide written informed consent obtained prior to participation in the study and any related procedures being performed
* Subjects willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examination.

Exclusion Criteria:

* Refusal of consent
* Women of childbearing potential without a negative pregnancy test; or women who are lactating.
* Any serious and/or unstable pre-existing medical disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acne who are actively considering enrolling in a clinical trial for said condition, but have not yet completed enrollment and randomization phases.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2026-06 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Rate of patients who decide to enroll in an acne clinical research. | 3 month
Number of acne study participants who remain in clinical study until completion. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Gill, Study Director — Power Life Sciences Inc.
Locations (1):
- Power Life Sciences, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Eichenfield DZ, Sprague J, Eichenfield LF. Management of Acne Vulgaris: A Review. JAMA. 2021 Nov 23;326(20):2055-2067. doi: 10.1001/jama.2021.17633. PMID 34812859
- [Background] Williams HC, Dellavalle RP, Garner S. Acne vulgaris. Lancet. 2012 Jan 28;379(9813):361-72. doi: 10.1016/S0140-6736(11)60321-8. Epub 2011 Aug 29. PMID 21880356
- [Background] Titus S, Hodge J. Diagnosis and treatment of acne. Am Fam Physician. 2012 Oct 15;86(8):734-40. PMID 23062156

DOCUMENTS (1):
  • Informed Consent Form (2025-05-30): https://cdn.clinicaltrials.gov/large-docs/58/NCT07010458/ICF_000.pdf